CLINICAL TRIAL: NCT04556695
Title: Exploration of Sedentary Behaviour Among General Practitioners: A Mixed Methods Study
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: University of Ulster (Other); University of Southern Denmark (Other); Loughborough University (Other)
Responsible Party: Principal Investigator, NeilHeron, Clinical Lecturer in GP, Queen's University, Belfast
Other Study IDs: MHLS 20_39 - Amendment 1
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Sedentary Behavior
Keywords: General Practitioner; Primary Care; Sedentary Behaviour; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Questionnaire survey: An initial online questionnaire, based on the International Sedentary Assessment Tool (ISAT), will be distributed to General Practice Specialty Trainees (GPSTs) and General Practitioners (GPs) throughout Northern Ireland.
  Interventions: Other: Questionnaire survey
- Accelerometer study: A purposive sample of questionnaire respondents will be asked to participate in the accelerometer study. This purposive sample will be based on responses to the online questionnaire. The aim will be to obtain a varied sample, based on questionnaire responses, by selecting individuals with a range of demographic characteristics and self-reported levels of sedentary behaviour. Some participants will also be asked to complete a further online survey, while wearing the accelerometer, regarding their health, wellbeing, burnout and fatigue.
  Interventions: Other: Questionnaire survey; Device: Accelerometer study
- Semi-structured interview study: A purposive sample comprising participants of the accelerometer study will be asked to participate in semi-structured interviews. This purposive sample will be based on the accelerometer data. The aim will be to obtain a varied sample, based on accelerometer data, by selecting individuals with a range of different levels of sedentary behaviour, demographic and workplace characteristics. The final number of participants will depend on the saturation of information.
  Interventions: Other: Questionnaire survey; Device: Accelerometer study; Other: Semi-structured interview study

INTERVENTIONS:
Other: Questionnaire survey — Online questionnaire, based on the International Sedentary Assessment Tool (ISAT)
Device: Accelerometer study — Consenting participants will be asked to wear an accelerometer on the lateral aspect of the middle of the right thigh (over the midpoint of the iliotibial band), continuously over a seven-day period.
  Groups: Accelerometer study; Semi-structured interview study
Other: Semi-structured interview study — Semi-structured interviews will take place via telephone or webcam. Participants will be given feedback regarding their accelerometer data relating to their levels of physical activity and sedentary behaviour. Questions will examine participants' thoughts and opinions regarding sedentary behaviour and physical activity in the General Practice setting. Further questions will explore participants' experiences of wearing accelerometers, their knowledge of and attitudes towards physical activity and sedentary behaviour and their thoughts or suggestions on interventions to reduce sedentary behaviour among GPs and GPSTs.
  Groups: Semi-structured interview study

SUMMARY:
A sequential, mixed-methods study exploring sedentary behaviour among General Practitioners and General Practice Specialty Trainees.

DETAILED DESCRIPTION:
The study follows a sequential, mixed-methods model involving three stages. The first stage will involve the dissemination of a questionnaire survey, in which participants will self-estimate their sedentary behaviour on a working day and on a non-working day. The second stage will involve the use of thigh-worn accelerometers and a sleep/work log to obtain objective data regarding sedentary behaviour among a purposive subset of participants who responded to the questionnaire. The third stage will involve semi-structured interviews with a purposive subset of participants who wore the accelerometers, which will be analysed with the application of a theoretical framework regarding the acceptability of healthcare interventions.

ELIGIBILITY:
Inclusion Criteria:

Participants will be General Practitioners or General Practice Specialty Trainees working in Northern Ireland, United Kingdom.

Exclusion Criteria:

Not working as a General Practitioner or General Practice Specialty Trainee in Northern Ireland, United Kingdom.

Min Age: 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General Practice Specialty Trainees (GPSTs) and General Practitioners (GPs) throughout Northern Ireland. GPs and GPSTs in Northern Ireland provide care for patients as part of the UK NHS, with working conditions similar to GPs and GPSTs throughout the rest of the UK.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Self-reported sedentary behaviour | Autumn 2020
Accelerometer measured sedentary behaviour | Autumn 2021
Thematic analysis of semi-structured interviews | Autumn 2021

CONTACTS AND LOCATIONS:
Overall Officials: Neil Heron, Principal Investigator — Centre for Public Health, Queen's University Belfast
Locations (1):
- Queen's University Belfast School of Medicine, Dentistry and Biomedical Sciences, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Sharing of study protocol to optimise openness and integrity of research.
Supporting Information: Study Protocol
Time Frame: Study protocol will be made available on commencement of the study and will be available for the duration of the study.
Access Criteria: Study protocol will be submitted for open access journal publication.